CLINICAL TRIAL: NCT03934736
Title: An Open-label, Single Arm Study, Evaluating the Immunogenicity and Safety of HEPLISAV-B® in Adults With End-Stage Renal Disease (ESRD) Undergoing Hemodialysis
Brief Title: HEPLISAV-B® in Adults With End-Stage Renal Disease (ESRD) Undergoing Hemodialysis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dynavax Technologies Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DV2-HBV-24
Record Dates: First submitted 2019-02-11; First posted 2019-05-02 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: End Stage Renal Disease on Hemodialysis (Diagnosis)
Keywords: ESRD; Hemodialysis; End Stage Renal Disease; Hepatitis B; HEPLISAV-B; Prevention and Control; HBV Vaccine; Hepatitis B Vaccine; HEPLISAV
MeSH Terms: conditions — Disease; Kidney Failure, Chronic; Hepatitis B | interventions — Heplisav-B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- HEPLISAV-B® (Experimental): A single dose of 0.5 mL HEPLISAV-B® administered intramuscularly in the deltoid muscle at Week 0 (Visit 1), Week 4 (Visit 2), Week 8 (Visit 3), and Week 16 (Visit 4).
  Interventions: Drug: HEPLISAV-B®

INTERVENTIONS:
Drug: HEPLISAV-B® — HEPLISAV-B®, a licensed, commercially-available hepatitis B vaccine for adults 18 years of age and older, consisting of the adjuvant cytidine phosphoguanosine (CpG) 1018 combined with the antigen recombinant hepatitis B surface antigen (rHBsAg).

SUMMARY:
This is an open-label, single arm study design to evaluate HEPLISAV-B® in adults with ESRD who are initiating or undergoing hemodialysis.

DETAILED DESCRIPTION:
Eligible participants will receive single doses of HEPLISAV-B® at Weeks 0, 4, 8, and 16 and will be followed through Week 68 or end of study (EOS). The study is designed to evaluate the immunogenicity over a 20-week period and safety over a 68-week period.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects at least 18 years of age
* Laboratory confirmed negative serology result to hepatitis B virus (HBV) surface antigen (HBsAg), antibody to hepatitis B surface antigen (anti-HBs), and antibody to hepatitis B core antigen (anti-HBc) prior to first study injection
* Must be clinically stable and in the opinion of the investigator able to comply with all study procedures
* Must be able and willing to provide informed consent
* Receiving hemodialysis or will initiate hemodialysis within 4 weeks of first study injection
* Women of childbearing potential (WOCBP) must consistently use an acceptable method of contraception or confirm in writing she will abstain from sexual activity from the Screening visit through 4 weeks after the last dose of study injection. Acceptable birth control methods include but are not limited to oral contraceptive medication, an intrauterine device (IUD), an injectable contraceptive (such as medroxyprogesterone acetate or Depo-Provera®), a birth control patch, or a barrier method (such as condom or diaphragm with spermicide).

Exclusion Criteria:

* Previous receipt of any hepatitis B vaccine
* History of human immunodeficiency virus (HIV) or hepatitis C virus (HCV) infection or antibody to HIV or HCV
* History of sensitivity to any component of study vaccine
* Substance or alcohol abuse that in the opinion of the investigator would interfere with compliance or with interpretation of the study results
* Recent or ongoing history of febrile illness (within 7 days of the first study injection)
* Has received any of the following prior to the first study injection:

  * Within 14 days:

    a. Any inactivated vaccine
  * Within 28 days:

    1. Systemic corticosteroids (more than 3 consecutive days) or other immunomodulatory or immune suppressive medication with the exception of inhaled steroids
    2. Any live virus vaccine
    3. Granulocyte colony-stimulating factor (G-CSF) or granulocyte-macrophage colony-stimulating factor (GM-CSF)
    4. Any other investigational medicinal agent
  * Within 90 days:

    1. Blood products or immunoglobulin
* If female and pregnant, nursing, or planning to become pregnant during the study
* Undergoing chemotherapy or expected to receive chemotherapy during the study period
* Has a medical condition considered by the investigator likely to interfere with the subject's compliance or the interpretation of study assessments, including the following laboratory abnormalities which the investigator may consider if severe:

  * Anemia
  * Thrombocytopenia
  * Leukocytosis
  * Neutropenia
  * Metabolic acidosis
  * Increased alanine aminotransferase (ALT) or aspartate aminotransferase (AST)
  * Hyperkalemia
  * Hypokalemia
* Is scheduled to undergo a kidney transplant within 6 months of the first study injection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2021-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Janssen, MD, Study Chair — Dynavax Technologies Corporation
Locations (20):
- United States (20):
  - DaVita Clinical Research or Affiliate, Bloomfield, Connecticut
  - DaVita Clinical Research or Affiliate, Middlebury, Connecticut
  - DaVita Clinical Research or Affiliate, Hollywood, Florida
  - DaVita Clinical Research or Affiliate, Ocala, Florida
  - DaVita Clinical Research or Affiliate, Tampa, Florida
  - DaVita Clinical Research or Affiliate, Winter Park, Florida
  - DaVita Clinical Research or Affiliate, Jeffersonville, Indiana
  - DaVita Clinical Research or Affiliate, Roseville, Michigan
  - DaVita Clinical Research or Affiliate, Edina, Minnesota
  - DaVita Clinical Research or Affiliate, Minneapolis, Minnesota
  - DaVita Clinical Research or Affiliate, Kansas City, Missouri
  - DaVita Clinical Research or Affiliate, Las Vegas, Nevada
  - DaVita Clinical Research or Affiliate, The Bronx, New York
  - DaVita Clinical Research or Affiliate, Asheville, North Carolina
  - DaVita Clinical Research or Affiliate, Canton, Ohio
  - DaVita Clinical Research or Affiliate, Philadelphia, Pennsylvania
  - DaVita Clinical Research or Affiliate, El Paso, Texas
  - DaVita Clinical Research or Affiliate, San Antonio, Texas
  - DaVita Clinical Research or Affiliate, Norfolk, Virginia
  - DaVita Clinical Research or Affiliate, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- HEPLISAV-B: A single dose of 0.5 mL HEPLISAV-B® administered intramuscularly in the deltoid muscle at Week 0 (Visit 1), Week 4 (Visit 2), Week 8 (Visit 3), and Week 16 (Visit 4).
  HEPLISAV-B®: HEPLISAV-B®, a licensed, commercially-available hepatitis B vaccine consisting of the adjuvant cytidine phosphoguanosine (CpG) 1018 combined with the antigen recombinant hepatitis B surface antigen (rHBsAg).
Period: Overall Study
Arm/Group | HEPLISAV-B
Started | 119
Completed | 86
Not Completed | 33

BASELINE CHARACTERISTICS:
Population: Enrolled Population
Groups:
- HEPLISAV-B®: A single dose of 0.5 mL HEPLISAV-B® administered intramuscularly in the deltoid muscle at Week 0 (Visit 1), Week 4 (Visit 2), Week 8 (Visit 3), and Week 16 (Visit 4).
  HEPLISAV-B®: HEPLISAV-B®, a licensed, commercially-available hepatitis B vaccine consisting of the adjuvant cytidine phosphoguanosine (CpG) 1018 combined with the antigen recombinant hepatitis B surface antigen (rHBsAg).
Arm/Group | HEPLISAV-B®
Number analyzed (Participants) | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (13.22)
Age, Continuous [Median (Full Range); unit: years] | 61.0 [22.0 to 87.0]
Age, Customized [Count of Participants; unit: Participants]
  18-55 | 47
  56+ | 72
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22
  Not Hispanic or Latino | 97
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 61
  White | 51
  More than one race | 7
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 119
Weight [Mean (Standard Deviation); unit: kg] | 89.9 (24.93)
Height [Mean (Standard Deviation); unit: cm] | 170.7 (10.39)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30.8 (8.14)
Smoking Status [Count of Participants; unit: Participants]
  Yes | 24
  No | 95
Diabetes Mellitus Status [Count of Participants; unit: Participants]
  Yes | 82
  No | 37
History of Hypertension [Count of Participants; unit: Participants]
  Yes | 116
  No | 3
Weight [Median (Full Range); unit: kg] | 89.2 [49.5 to 182.3]
Height [Median (Full Range); unit: cm] | 170.2 [137.2 to 195.6]
Body Mass Index [Median (Full Range); unit: kg/m^2] | 30.1 [18.3 to 57.6]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Reporting Clinically Significant Adverse Events - Medically-attended Adverse Events, Serious Adverse Events, and Immune-mediated Adverse Events of Special Interest
Description: Proportion of participants with Medically-attended adverse events (MAEs), Serious Adverse Events (SAEs), and immune-mediated Adverse Events of Special Interest (AESIs). MAEs are Adverse events (AEs) for which a subject sought medical attention at a doctor's office, clinic or study site, or emergency room, or was hospitalized. SAEs are AEs that met the definition of Serious per FDA regulations.
Time Frame: Week 0 (Visit 1) until Week 68 or early termination
Population: Safety Population: All participants who received at least 1 study injection and who had any post-baseline safety data
Measure: Number; unit: percentage of participants
Arm/Group | HEPLISAV-B
Number analyzed (Participants) | 119
percentage of participants
  New-onset Immune-mediated Adverse Events | 0.8
  Medically-attended Adverse Events | 66.4
  Serious Adverse Events | 48.7

2. Primary Outcome: Seroprotection Rate (SPR) = Percentage of Participants Who Have a Seroprotective Immune Response
Description: SPR is the percentage of participants who have a seroprotective immune response (antibody level to anti-HBsAg greater than or equal to 10 milli-international unit [mIU]/mL) after HEPLISAV-B
Time Frame: Week 20
Population: Per protocol subjects at Week 20
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HEPLISAV-B®
Number analyzed (Participants) | 75
percentage of participants | 89.3 [80.1 to 95.3]

3. Secondary Outcome: Percentage of Subjects With Anti-HBs Concentration ≥100 mIU/mL
Description: Percentage of subjects with anti-HBs concentration ≥100 mIU/mL.
Time Frame: Weeks 4, 8, 16, 20
Population: Per protocol subjects at Weeks 4, 8,16, 20
Measure: Number (95% Confidence Interval); unit: percentage of subjects with anti-HBs≥100
Arm/Group | HEPLISAV-B
Number analyzed (Participants) | 75
percentage of subjects with anti-HBs≥100
  Week 4: number analyzed (Participants) | 74
  Week 4 | 5.4 [1.5 to 13.3]
  Week 8: number analyzed (Participants) | 74
  Week 8 | 33.8 [23.2 to 45.7]
  Week 16 | 57.3 [45.4 to 68.7]
  Week 20 | 81.3 [70.7 to 89.4]

4. Secondary Outcome: Serum Anti-HBsAg Geometric Mean Concentration (GMC)
Description: Serum Anti-HBsAg Geometric Mean Concentration (GMC).
Time Frame: Weeks 4, 8, 16, 20
Population: Per protocol subjects at Week 4, 8, 16, 20
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | HEPLISAV-B
Number analyzed (Participants) | 75
mIU/mL
  Week 4: number analyzed (Participants) | 74
  Week 4 | 4.4 [3.0 to 6.5]
  Week 8: number analyzed (Participants) | 74
  Week 8 | 33.5 [17.5 to 64.3]
  Week 16 | 155.3 [81.5 to 296.2]
  Week 20 | 1061.8 [547.2 to 2060.2]

5. Secondary Outcome: Seroprotection Rate (SPR) = Percentage of Participants Who Have a Seroprotective Immune Response
Description: as for outcome 2
Time Frame: Weeks 4, 8, 16, 20
Population: Per protocol subjects at Weeks 4, 8,16, 20
Measure: Number (95% Confidence Interval); unit: SPR percent (≥ 10 mIU/mL)
Arm/Group | HEPLISAV-B
Number analyzed (Participants) | 75
SPR percent (≥ 10 mIU/mL)
  Week 4 | 20.3 [11.8 to 31.2]
  Week 8 | 56.8 [44.7 to 68.2]
  Week 16 | 78.7 [67.7 to 87.3]
  Week 20 | 89.3 [80.1 to 95.3]

ADVERSE EVENTS:
Time Frame: The reporting period for All-Cause Mortality, Serious Adverse Events, and Other (Not Including Serious) Adverse Events begins at the time of the first study treatment from Visit 1 (Week 0) through EOS Visit (Week 68).
Description: An MAE is an AE for which a subject sought medical attention at a doctor's office, clinic, study site, emergency room, or was hospitalized. In this trial, only MAEs were collected. Medical conditions present at Screening (ie, before informed consent was obtained) or present before the first study treatment (Day 1) are medical history, not MAEs. Any increase in severity or frequency of a medical condition documented as medical history after the first study treatment was recorded as an MAE
Arm/Group | HEPLISAV-B
All-Cause Mortality (participants affected / at risk) | 14/119
Serious Adverse Events (participants affected / at risk) | 58/119
Other Adverse Events (participants affected / at risk) | 0/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HEPLISAV-B (N=119)
Anemia (Blood and lymphatic system disorders) | 5
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Acute Left Ventricular Failure (Cardiac disorders) | 1
Acute Myocardial Infarction (Cardiac disorders) | 3
Angina Pectoris (Cardiac disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 2
Bradycardia (Cardiac disorders) | 2
Cardiac Arrest (Cardiac disorders) | 2
Cardiac Failure (Cardiac disorders) | 2
Cardiac Failure Acute (Cardiac disorders) | 1
Cardiac Failure Congestive (Cardiac disorders) | 2
Cardiogenic Shock (Cardiac disorders) | 1
Coronary Artery Stenosis (Cardiac disorders) | 1
Mitral Valve Incompetence (Cardiac disorders) | 1
Sickle Cell Anaemia (Congenital, familial and genetic disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Gastric Antral Vascular Ectasia (Gastrointestinal disorders) | 1
Gastric Polyps (Gastrointestinal disorders) | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 5
Haematemesis (Gastrointestinal disorders) | 2
Impaired Gastric Emptying (Gastrointestinal disorders) | 1
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 3
Melaena (Gastrointestinal disorders) | 1
Oesophageal Food Impaction (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Pancreatitis Acute (Gastrointestinal disorders) | 1
Pancreatitis Chronic (Gastrointestinal disorders) | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 1
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1
Chest Discomfort (General disorders) | 1
Death (General disorders) | 2
Gait Disturbance (General disorders) | 1
Non-Cardiac Chest Pain (General disorders) | 1
Pyrexia (General disorders) | 2
Cholecystitis (Hepatobiliary disorders) | 1
Hepatotoxicity (Hepatobiliary disorders) | 1
Abdominal Abscess (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 4
Clostridium Difficile Colitis (Infections and infestations) | 2
Clostridium Difficile Infection (Infections and infestations) | 1
Corona Virus Infection (Infections and infestations) | 4
Diverticulitis (Infections and infestations) | 3
Epididymitis (Infections and infestations) | 1
Gangrene (Infections and infestations) | 2
Influenza (Infections and infestations) | 1
Localised Infection (Infections and infestations) | 2
Oesophageal Candidiasis (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 2
Osteomyelitis Chronic (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 9
Pneumonia Viral (Infections and infestations) | 3
Pyelonephritis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 5
Septic Shock (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 2
Urosepsis (Infections and infestations) | 1
Acetabulum Fracture (Injury, poisoning and procedural complications) | 1
Arteriovenous Fistula Site Haemorrhage (Injury, poisoning and procedural complications) | 1
Exposure to Household Chemicals (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Intentional Overdose (Injury, poisoning and procedural complications) | 1
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1
Rib Fracture (Injury, poisoning and procedural complications) | 1
Anticoagulation Drug Level Above Therapeutic (Investigations) | 2
Blood Culture Positive (Investigations) | 1
Coronavirus Test Positive (Investigations) | 2
Acidosis (Metabolism and nutrition disorders) | 1
Adult Failure to Thrive (Metabolism and nutrition disorders) | 1
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 2
Electrolyte Imbalance (Metabolism and nutrition disorders) | 1
Fluid Overload (Metabolism and nutrition disorders) | 4
Gout (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Ketosis (Metabolism and nutrition disorders) | 1
Lactic Acidosis (Metabolism and nutrition disorders) | 1
Metabolic Acidosis (Metabolism and nutrition disorders) | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1
Brain Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Papillary Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral Haemorrhage (Nervous system disorders) | 1
Metabolic Encephalopathy (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 4
Device Damage (Product Issues) | 1
Device Malfunction (Product Issues) | 1
Azotaemia (Renal and urinary disorders) | 2
End Stage Renal Disease (Renal and urinary disorders) | 2
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 4
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1
Hidradenitis (Skin and subcutaneous tissue disorders) | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1
Aortic Stenosis (Vascular disorders) | 1
Aortitis (Vascular disorders) | 1
Hypertensive Emergency (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2
Temporal Arteritis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no multicenter publication has occurred within 18 months of the completion of this Study, Investigator shall have the right to publish or present independently the results of this Study. Investigator shall provide Dynavax with a copy of any such presentation/publication derived from the Study for review at least 30 days in advance of submission. Except for the Study Data, Dynavax reserves the right to delete any Intellectual Property or other confidential information of Dynavax.

DOCUMENTS (2):
  • Study Protocol (2020-04-17): https://cdn.clinicaltrials.gov/large-docs/36/NCT03934736/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-15): https://cdn.clinicaltrials.gov/large-docs/36/NCT03934736/SAP_001.pdf